CLINICAL TRIAL: NCT07400003
Title: A Randomized, Double-Blind, Controlled Phase I/II Clinical Trial to Evaluate the Safety and Immunogenicity of Different Doses of a Lyophilized Herpes Zoster Virus mRNA Vaccine in Adults Aged 40 Years and Older
Brief Title: Study to Evaluate the Safety and Immunogenicity of a Lyophilized Herpes Zoster Virus mRNA Vaccine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-mHZ-1001
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Herpes Zoster; mRNA Vaccine
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-dose group (Experimental): Participants will receive two doses of lyophilized herpes zoster virus mRNA vaccine (low dosage), with 30 days or 60 days apart
  Interventions: Biological: Low-dose experimental vaccine
- High-dose group (Experimental): Participants will receive two doses of lyophilized herpes zoster virus mRNA vaccine (high dosage), with 30 days or 60 days apart
  Interventions: Biological: High-dose experimental vaccine
- Comparator A (Active Comparator): Participants will receive a single dose of saline on day 0 and a single dose of herpes zoster vaccine, live on day 60
  Interventions: Biological: Active-controlled vaccine A
- Comparator B (Active Comparator): Participants will receive two doses of recombinant zoster vaccine (CHO cell), with 60 days apart
  Interventions: Biological: Active-controlled vaccine B
- Comparator C (Placebo Comparator): Participants will receive two doses of saline, with 60 days apart
  Interventions: Other: Placebo group

INTERVENTIONS:
Biological: Low-dose experimental vaccine — Lyophilized herpes zoster virus mRNA vaccine
  Arms: Low-dose group
Biological: High-dose experimental vaccine — Lyophilized herpes zoster virus mRNA vaccine
  Arms: High-dose group
Biological: Active-controlled vaccine A — herpes zoster attenuated live vaccine, lyophilized
  Arms: Comparator A
Biological: Active-controlled vaccine B — Shingrix®
  Arms: Comparator B
Other: Placebo group — Saline
  Arms: Comparator C

SUMMARY:
This clinical trial included two parts, Part A and Part B. The goal of Part A is to evaluate the safety and preliminary immunogenicity of the lyophilized herpes zoster virus mRNA vaccine (HZ mRNA vaccine) in healthy populations aged 40 years and older. The goal of Part B is to select the optimal dosage and schedule in healthy populations aged 50 years and older to support next further study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, controlled study. Part A employed sequential enrollment by age and dosage. All participants received two doses of the study vaccine. Safety observation conducted throughout the study. Humoral and celluar immunity were evaluated.

In Part B, participants randomly received either different dosage study vaccine or active controlled vaccine, with different immunization schedule. Safety observation conducted throughout the study. Humoral and celluar immunity were evaluated. Immune persistence was also evaluated at multiple timepoints after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Age ≥ 40 years; Phase II: Age ≥ 50 years;
* Participants are able to understand and voluntarily sign the informed consent form;
* Able to provide legal identification;
* Participants of childbearing potential and their sexual partners agree to voluntarily adopt effective contraceptive measures from the signing of the informed consent form until 6 months after the last dose of the investigational vaccine, with no plans for sperm or egg donation;
* Agree to comply with the visit schedule, sample collection, vaccination, and other trial procedures throughout the study period, and remain accessible at all times during the trial.

Exclusion Criteria:

* History of chickenpox or herpes zoster in adulthood;
* History of chickenpox or herpes zoster vaccination (including administration of registered products or participation in clinical trials of chickenpox or herpes zoster vaccines);
* Close contact with patients infected with chickenpox or herpes zoster within the past 30 days;
* Clinically significant abnormalities in protocol-specified clinical laboratory tests prior to vaccination (applicable to Phase I clinical trials only):

A. Hematological parameters: White blood cell count (WBC), hemoglobin (Hb), platelet count (Plt); B. Blood biochemical parameters: Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), fasting blood glucose (Glu), creatinine (CR); C. Urinalysis parameter: Urine protein (PRO); D. Coagulation parameters: Prothrombin time (PT), activated partial thromboplastin time (APTT), fibrinogen (Fib), international normalized ratio (INR); E. 12-lead electrocardiogram (ECG).

* Poorly controlled chronic diseases or significant medical history, including but not limited to cardiovascular diseases (e.g., poorly controlled hypertension defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg for participants aged 40-59 years prior to enrollment, or systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg for participants aged ≥60 years), metabolic disorders (e.g., poorly controlled diabetes), hematological diseases, hepatic or renal diseases, digestive system diseases, respiratory system diseases, history of major organ transplantation, or malignancy within the past five years;
* History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or any condition that increases the risk of myocarditis or pericarditis;
* Autoimmune diseases, immunodeficiency diseases, or family history thereof (including but not limited to psoriasis, systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid diseases, acute disseminated encephalomyelitis, facial paralysis, hypersensitivity reactions, polymyalgia rheumatica, rheumatoid arthritis, Guillain-Barré syndrome, asplenia, functional asplenia, HIV infection);
* Coagulation disorders (e.g., coagulation factor deficiencies, platelet abnormalities, or other coagulopathies);
* Current or previous severe neurological disorders (epilepsy, convulsions, or seizures) or psychiatric illnesses, or family history of psychiatric disorders;
* Acute illnesses or acute exacerbations of chronic diseases within the past 7 days, or known or suspected active infections;
* Immunosuppressive therapy or other immunomodulatory treatments (prednisone ≥20 mg/day or equivalent for >14 days), cytotoxic therapy within the past 6 months, or planned use during the trial;
* Administration of immunoglobulins or other blood products within the past 3 months (use of hepatitis B immunoglobulin within the past 1 month), or planned use during the trial;
* Participation in other clinical studies within the past 30 days or planned participation during this trial;
* Vaccination with live-attenuated vaccines or nucleic acid vaccines within the past 28 days, or vaccination with subunit, inactivated, or other types of vaccines within the past 14 days;
* Known allergy to vaccines or vaccine components, such as urticaria, dyspnea, or angioedema following vaccination;
* Pregnancy, lactation, or positive urine pregnancy test in female participants;
* Fever (axillary temperature ≥37.3°C) within 3 days prior to vaccination or use of antipyretics, analgesics, or antihistamines (e.g., acetaminophen, ibuprofen, loratadine, cetirizine, etc.) as reported during inquiry;
* Physical examination deemed unsatisfactory on the day of planned vaccination;
* Skin lesions, inflammation, ulcers, rashes, scars, or other conditions at the target injection site that may interfere with administration or local reaction assessment;
* Any other factors deemed by the investigator to render the participant unsuitable for participation in the clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 519 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse reactions within 30 days | 0~30 days after each dose vaccination
  The incidence of adverse reactions within 0~30 days after each dose vaccination.
Seroconversion rate of gE antibody | Day 30 after two doses
  The seroconversion rate of gE antibody on Day 30 after two doses vaccination.
Geometric mean concentration (GMC) of gE antibody | Day 30 after two doses
  The GMC of gE antibody on Day 30 after two doses vaccination.

SECONDARY OUTCOMES:
Adverse reactions within 0~14 days | 0~14 days after each dose vaccination
  The incidence of adverse reactions within 0~14 days after each dose vaccination.
Incidence of serious adverse events (SAEs) | From the first dose to 12 months after the second dose
  The incidence of SAEs from the first dose to 12 months after the second dose.
Incidence of adverse events of special interest（AESI) | From the first dose to 12 months after the second dose
  The incidence of AESI from the first dose to 12 months after the second dose.
GMC of gE antibody | On Day 30 or Day 60 after the first dose, and on Day 14、Day 180 and Day 360 after the second dose
  The GMC of gE antibody on Day 30 or Day 60 after the first dose, and on Day 14、Day 180 and Day 360 after the second dose
Geometric mean fold rise (GMFR) of gE antibody | On Day 30 or Day 60 after the first dose, and on Day 14 and Day 30 after the second dose
  The GMFR of gE antibody on Day 30 or Day 60 after the first dose, and on Day 14 and Day 30 after the second dose
Seroconversion rate of varicella-zoster virus (VZV) antibody | On Day 30 or Day 60 after the first dose, and on Day 14、Day 30、Day 180 and Day 360 after the second dose
  The seroconversion rate of VZV antibody on Day 30 or Day 60 after the first dose, and on Day 14、Day 30、Day 180 and Day 360 after the second dose.
GMT of VZV antibody | On Day 30 or Day 60 after the first dose, and on Day 14、Day 30、Day 180 and Day 360 after the second dose
  The GMT of VZV antibody on Day 30 or Day 60 after the first dose, and on Day 14、Day 30、Day 180 and Day 360 after the second dose
GMFR of VZV antibody | On Day 30 or Day 60 after the first dose, and on Day 14 and Day 30 after the second dose
  The GMFR of VZV antibody on Day 30 or Day 60 after the first dose, and on Day 14 and Day 30 after the second dose
Frequency of CD4/CD8+ T cells secreting gE-specific cytokines | On Day 30 or Day 60 after the first dose, and on Day 14、Day 30、Day 180 and Day 360 after the second dose
  The frequency of CD4/CD8+ T cells secreting gE-specific cytokines (IFN-γ, IL-2, TNF-α, CD40L) on Day 30 or Day 60 after the first dose, and on Day 14、Day 30、Day 180 and Day 360 after the second dose.
Cellular immune response rate | On Day 30 or Day 60 after the first dose, and on Day 14 and Day 30 after the second dose
  The cellular immune response rate on Day 30 or Day 60 after the first dose, and on Day 14 and Day 30 after the second dose.

CONTACTS AND LOCATIONS:
Overall Officials: Na Xie, Principal Investigator — Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention
Locations (1):
- Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No